CLINICAL TRIAL: NCT01181063
Title: Pharmacokinetic Pilot Study on Budesonide/Formoterol Easyhalers and Symbicort Turbuhaler; an Open, Randomised, Single Centre, Single Dose Study With Crossover Design in Healthy Subjects
Brief Title: Pharmacokinetic Pilot Study on Budesonide/Formoterol Device-metered Dry Powder Inhalers
Acronym: Reco-Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Irja Korpela, Clinical Study Director, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3103005
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Asthma; Easyhaler
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Nebulizers and Vaporizers; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 400/12 μg D94-2BF (60/40) inhaler (Experimental)
  Interventions: Drug: Budesonide/formoterol 320/9 μg and 400/12 μg inhalers
- 320/9 μg D94-2BF (20/80) inhaler (Experimental)
  Interventions: Drug: Budesonide/formoterol 320/9 μg and 400/12 μg inhalers
- Symbicort 320/9 μg inhaler (Active Comparator)
  Interventions: Drug: Budesonide/formoterol 320/9 μg and 400/12 μg inhalers
- 320/9 μg D94-2F (60/40) inhaler (Experimental)
  Interventions: Drug: Budesonide/formoterol 320/9 μg and 400/12 μg inhalers
- 320/9 μg D94-2BF (60/40) inhaler (Experimental)
  Interventions: Drug: Budesonide/formoterol 320/9 μg and 400/12 μg inhalers

INTERVENTIONS:
Drug: Budesonide/formoterol 320/9 μg and 400/12 μg inhalers — Budesonide/formoterol 320/9 μg and 400/12 μg in different kind of inhalers and Symbicort Turbuhaler forte 320/9 μg. Ech subject will be randomly allocation to 4 of 5 products, a single dose administration of each product
  Other Names: Symbicort 320/9 μg inhaler

SUMMARY:
Due to the complexity of orally inhaled products (combination of a formulation and a device)and the topical nature of drug delivery to the lung for efficacy in vitro-in vivo correlation(IVIVC) for inhaled dosage forms is not generally known.

The rationale of this pilot study is to gain in vivo data of the Budesonide/formoterol EH product variants under development and compare pulmonary deposition (administration with charcoal) of different product variants of Budesonide/formoterol EH with Symbicort TH.

DETAILED DESCRIPTION:
In order to reduce variability, a crossover design is chosen. An open study design is regarded appropriate because the study is a pilot and the primary study variables are pharmacokinetic(PK) parameters derived from drug concentrations in plasma. Wash-out period of at least 3 days between the study treatment administration days is considered sufficient for the elimination of budesonide and formoterol.

The single dose study is suitable for this kind of study, where the aim is to compare products and the therapeutic response is not measured.

The dose level selected is 2 inhalations (single dose) for all products. The administration of 2 inhalations enables the determination of budesonide and formoterol concentrations in plasma.

In this study the investigational products are administered concomitantly with oral charcoal to block the GI absorption and to assess the pulmonary deposition of the active substances.

Comparison of pulmonary deposition between the products is considered more relevant than systemic exposure at this point of product development. In the pivotal PK study total systemic exposure will also be assessed.

Blood samples for formoterol analysis will be collected up to 24 hours and for budesonide analysis up to 12 hours after dosing to cover at least 80% of the total area under the concentration-time curve from time zero extrapolated to infinity (AUC∞).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history, and laboratory and physical examinations.
* Finnish speaking males and females, 18-60 (inclusive) years of age.
* Normal weight defined as body mass index (BMI) > 19 and < 30 kg/m2 (BMI = weight/height2)
* Weight at least 50 kg
* Hemoglobin 135-195 g/l male, 125-175 g/l female.

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study.
* Intake of any medication that could affect the outcome of the study. As an exception, contraceptives and hormone replacement therapy are allowed.
* Any clinically significant abnormal laboratory value or physical finding (including electrocardiogram [ECG] and vital signs) that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study, as judged by the investigator.
* Known hypersensitivity to the active substance(s) or to any of the excipients of the drug.
* History of vasovagal collapses.
* History of anaphylactic/anaphylactoid reactions.
* History of seizures including febrile seizures.
* Pregnant or lactating females.
* Females of childbearing potential not using proper contraception (mechanical and/or hormonal contraception, intrauterine device [IUD] or surgical sterilization) Note: Females of childbearing potential with no current sexual relationship can be included without contraception according to the judgement of the investigator.
* Recent or current (suspected) drug abuse or positive result in the drugs abuse test.
* Recent or current alcohol abuse (regular drinking more than 21 units per week for males and more than 16 units per week for females [1 unit = 4 cl spirits or equivalent]).
* Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the study(from the screening visit to the end-of study visit).
* Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from the use of caffeine containing beverages during the treatment periods until 24h after study treatment administration.
* Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration.
* Administration of another investigational drug within 90 days prior to the first study treatment administration.
* Unsuitable veins for repeated venipuncture or for cannulation.
* Inability to learn the correct inhalation technique (during screening or on a separate visit for training).
* Predictable poor compliance or inability to communicate well with the study centre personnel.
* Inability to participate in all treatment periods.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The maximum observed concentration of concentration-time curve. | 24 hours

SECONDARY OUTCOMES:
The area under the concentration-time curve from time zero to infinity, AUC∞ | 24 hours
  The area under the concentration-time curve from time zero to infinity will be determined by adding AUCt to the extrapolated area that will be determined dividing the last quantifiable concentration by terminal elimination rate constant from log-linear portion of a concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Ingman, MD, PhD, Principal Investigator — Phase I Unit, Orion Pharma, Espoo, Finland
Locations (1):
- Phase I Unit, Orion Pharma, Espoo, Finland